CLINICAL TRIAL: NCT06366581
Title: Transcriptomic Analysis of Incisional Hernia Based on High-throughput Sequencing Technology
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Other Study IDs: HD20240307
Record Dates: First submitted 2024-03-07; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Incisional Hernia; Extracellular Matrix Alteration
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IH group: Patients who underwent incisional hernia repair were defined as the experimental group (labelled as the IH group)
  Interventions: Diagnostic Test: Transcriptomic analysis
- NC group: patients who underwent laparoscopic cholecystectomy were defined as the control group (labelled as the NC group)
  Interventions: Diagnostic Test: Transcriptomic analysis

INTERVENTIONS:
Diagnostic Test: Transcriptomic analysis — high-throughput sequencing technology

SUMMARY:
This study included patients who underwent surgical treatment for incisional hernia and non-hernia conditions. Surgical specimens were collected for transcriptome sequencing to obtain the gene expression list. Then genes analyzed by Gene Ontology, protein interactions, and signaling pathway enrichment using the expression matrix.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 75 years 2.diagnosed with incisional hernia 3.normal tumour markers 4.elective surgery patients.

Exclusion Criteria:

1. patients with vital organ failure (heart liver, lung, kidney and others)
2. malignant tumors not been completely relieved by active treatment,
3. patients who have psychiatric diseases or comprehension disorders.
4. patients with metabolic disease involving connective tissue collagen.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent incisional hernia repair were defined as the experimental group (labelled as the IH group), and patients who underwent laparoscopic cholecystectomy were defined as the control group (labelled as the NC group).
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
the gene expression list | 2023.3-2023.9
  the gene expression list

CONTACTS AND LOCATIONS:
Locations (1):
- Hua Dong Hospital Affiliated to Fu Dan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided